CLINICAL TRIAL: NCT04729348
Title: Phase II Trial of Pembrolizumab and Lenvatinib for Leptomeningeal Metastases
Brief Title: Pembrolizumab And Lenvatinib In Leptomeningeal Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Planned interim analysis
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Nancy Wang, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-533
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor; Solid Tumor, Adult; Leptomeningeal Metastasis
Keywords: Solid Tumor; Solid Tumor, Adult; Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PEMBROLIZUMAB and LENVATINIB (Experimental): The research study procedures include screening for eligibility and study treatment, including evaluations and follow up visits.
  * PEMBROLIZUMAB daily, every 3 weeks
  * LENVATINIB daily every 3 weeks
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — Oral, daily, dosage per protocol
  Other Names: Keytruda®
Drug: Lenvatinib — Oral, daily, dosage per protocol
  Other Names: Lenvima™

SUMMARY:
The purpose of this research is to examine if an experimental drug combination impacts the survival rate of individuals with Leptomeningeal Metastases

This research study involves an experimental drug combination.

The names of the study drugs involved in this study are:

* Pembrolizumab
* Lenvatinib

DETAILED DESCRIPTION:
This is a single arm Phase 2 study of pembrolizumab in combination with lenvatinib in patients with leptomeningeal metastases from any solid tumor.

The research study procedures include screening for eligibility and study treatment, including evaluations and follow up visits.

* The names of the study drugs involved in this study are:
* Pembrolizumab
* Lenvatinib

The study treatment will last for up to 35 cycles (a cycle is 21 days long), or until the disease gets worse or unacceptable side effects. Participants will be followed for up to 90 days after the end of the study treatment.

It is expected that about 19 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug combination to learn whether the drug combination works in treating a specific disease. "Investigational" means that the drug combination is being studied.

The U.S. Food and Drug Administration (FDA) has not approved pembrolizumab or lenvatinib for this specific disease but each has been approved for other uses.

.

.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed solid malignancy.
* Leptomeningeal metastases, as determined by: 1) positive CSF cytology, or 2) MRI suggestive of leptomeningeal metastases and atypical cytology.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of pembrolizumab in combination with lenvatinib in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status ≤ 1 (Karnofsky ≥70%, see Appendix A)
* Participants must have normal organ and marrow function; all screening labs should be performed within 14 days of treatment initiation.
* Eligibility Criteria for Organ and Marrow Function

  * Hematological

    * Absolute neutrophil count (ANC) ≥1500/μL
    * Platelets ≥100 000/μL
    * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La
  * Renal

    --- Creatinine ≤1.5 × ULN OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
  * Hepatic

    * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
    * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
  * Coagulation

    * International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Female participants of childbearing potential should have a negative urine pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* A female participant is eligible to participate if she is not pregnant not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study medication
* A male participant must agree to use a contraception as detailed in this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
* If participant is on a daily steroid medication, dose must be stable at ≤2 mg dexamethasone (or equivalent) for 7 days prior to initiation of treatment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have received prior systemic anti-cancer therapy including investigational agents within 14 days of protocol treatment. Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Participant must have recovered adequately from the toxicity and/or complications from any prior surgical procedures prior to starting therapy. Lenvatinib should be held for 4 weeks following a major surgical procedure, 2 weeks following a minor surgical procedure.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pembrolizumab. In addition, these participants are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated. No testing for HIV, Hepatitis B, and Hepatitis C is required unless mandated by local health authority.
* Participants who are receiving any other investigational agents.
* Has a diagnosis of immunodeficiency.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known additional malignancy that is progressing or requires active treatment (except for patients receiving letrozole, anastrozole, exemestane, tamoxifen, fulvestrant, trastuzumab, bisphosphonates, denosumab or ovarian suppression therapy). Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of system.
* Requires treatment with high dose systemic corticosteroids defined as dexamethasone >2mg/day or bioequivalent within 7 days of initiating therapy.
* Has received systemic immunosuppressive treatments, aside from systemic corticosteroids as described in Section 3.2.15, within three months of start of study drug.
* Severe hypersensitivity (Grade 3 or higher) to pembrolizumab, lenvatinib, or any of their excipients.
* Has received prior treatment with any treatment targeting VEGF-directed angiogenesis, any anti-PD-1, anti-PD-L1, anti-PD-L2 agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Has a known history of active TB (Bacillus Tuberculosis).
* Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study treatment.
* Bleeding or thrombotic disorders or participants at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels (e.g., carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
* Participants having > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
* Uncontrolled hypertension (Systolic BP>140 mmHg or diastolic BP >90 mmHg) in spite of an optimized regimen of antihypertensive medication.
* Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
* Prolongation of corrected QT (QTc) interval to >480 milliseconds (ms).
* Serious nonhealing wound, ulcer, or bone fracture.
* Has had an allogenic tissue/solid organ transplant (large organ transplants, stem-cell transplant requiring chronic immunosuppressant therapy necessary to prevent graft rejection).
* Will need immediate local surgery or radiation for brain metastases.
* Unable to undergo MRI.
* Electrolyte abnormalities that have not been corrected.
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants alive at 6 months | 6 months
  The proportion of patients alive at 6 months will be summarized with a 90% confidence interval estimated using the method of Atkinson and Brown (Biometrics, 1985), which allows for the two-stage design. Based on a sample of 19 patients, the confidence interval will be no wider than 33%

SECONDARY OUTCOMES:
Proportion of Participants with Grade 3 or higher toxicities | first dose of study treatment up to the 30-Day Post Drug Visit up to 30 Months
  The proportion of patients with Grade 3 or higher toxicities will be presented with 90% exact binomial confidence intervals. The incidence of events that are new or worsening from the time of first dose of treatment will be summarized according to system organ class and/or preferred term, severity (based on Common Terminology Criteria for Adverse Events v5.0 CTCAE grade), type of adverse event, and relation to study treatment. Deaths reportable as SAEs and non-fatal serious adverse events will be listed by patient and tabulated by primary system organ class, and type of adverse event
Proportion of evaluable participants with intracranial/intraspinal response | 30 Months
  The proportion of evaluable patients with intracranial/intraspinal response (CR or PR by RANO) will be presented with a two-sided, 90% exact binomial confidence interval.
Proportion of evaluable participants with extracranial response | 30 Months
  The proportion of evaluable patients with extracranial response (CR or PR by RECIST 1.1) will be presented with a two-sided, 90% exact binomial confidence interval.
  For a sample of 19 patients, the confidence interval will have maximum width of 33%
Intracranial/intraspinal Progression Free Survival (IPFS) | 30 Months
  The distribution of intracranial/intraspinal PFS (IPFS) in participants will be summarized using the method of Kaplan-Meier. IPFS is defined as the time from registration to documented intracranial/intraspinal progression (RANO) or death, whichever occurs first.
  Patients who have neither died nor progressed at the time of analysis will be censored at the date of last adequate disease assessment.
Median Intracranial/intraspinal Progression Free Survival (IPFS) | 30 Months
  Median IPFS will be presented and accompanied by 90% confidence intervals estimated using log(-log(survival)) methodology. Point estimates at 3 and 6 months will also be presented with confidence intervals.
  .
Extracranial Progression Free Survival (EPFS) | 30 Months
  The distribution of extracranial PFS (EPFS) will be summarized using the method of Kaplan-Meier. EPFS is defined as the time from registration to documented extracranial progression (RANO) or death, whichever occurs first. Patients who have neither died nor progressed at the time of analysis will be censored at the date of last adequate disease assessment.
Median Extracranial Progression Free Survival (EPFS) | 30 Months
  Median EPFS will be presented and accompanied by 90% confidence intervals estimated using log(-log(survival)) methodology. Point estimates at 3 and 6 months will also be presented with confidence intervals.
Overall Survival | 30 Months
  The distribution of overall survival will be summarized using the method of Kaplan-Meier. (OS) is defined as the time from registration to death due to any cause, or censored at date last known alive
Median Overall Survival | 30 Months
  median OS will be presented and accompanied by 90% confidence intervals estimated using log(-log(survival)) methodology. (OS) is defined as the time from registration to death due to any cause, or censored at date last known alive
Proportion of participants with leptomeningeal metastases from breast cancer alive | 6 months
  The proportion of patients with leptomeningeal metastases from breast cancer alive at 6 months will be summarized with a 90% two-sided, exact binomial confidence interval. The maximum width of the confidence intervals is 0.55.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Wang, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation